CLINICAL TRIAL: NCT00769717
Title: Comparative Health Improvements and Rate of Relapse in Weight-Centered vs. Wellness-Centered Interventions for Obese Women
Brief Title: Evaluation of a Health at Every Size vs a Behavioral Weight Loss Approach for Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Reading Hospital and Medical Center (Other)
Collaborators: The Edna G. Kynett Memorial Foundation (Other)
Responsible Party: Principal Investigator, Janell Mensinger, PhD, FAED, Associate Research Professor, Villanova University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRHMC 02708
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: obesity; wellness; cardiovascular disease prevention; health at every size; weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: 1:1 Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There was full allocation concealment through the 3-month recruitment phase of the trial.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wellness-Centered (Experimental): A health at every size intervention, the HUGS program was conceived and developed in 1987 by Linda Omichinski, Registered Dietitian. HUGS stands for Health focused, Understanding lifestyle, Group supported, and Self-esteem building. It is an integrated approach that promotes healthy eating, active living, and self acceptance regardless of weight. HUGS teaches strategies to recognize and respond to physiological signs of hunger and satiety to determine food intake. The manualized curriculum is accompanied by the books Tailoring Your Tastes and Staying Off of the Diet Roller Coaster which participants will receive in addition to a booklet of handouts. Kelly Bliss, a psychotherapist and fitness professional with 17 years experience in health-centered approaches for weight management, will deliver the intervention in 2 groups of 20 people that meet weekly for 6 months.
  Interventions: Behavioral: Wellness-Centered (HUGS)
- Weight-Centered (Active Comparator): The LEARN Program for Weight Management is an evidence-based behavior modification approach to weight loss developed by Dr. Kelly Brownell, Ph.D. Psychologist. LEARN is an acronym that stands for Lifestyle, Exercise, Attitudes, Relationships, and Nutrition. This manualized curriculum shares many principals with the HUGS program in that both emphasize the importance of healthy lifestyle choices and gradual sustainable change. However, the LEARN program makes weight loss an explicit goal and focuses more on food intake levels based on external prescriptions and caloric restriction. Participants in the LEARN program will receive the LEARN Program for Weight Management manual and the LEARN Weight Stabilization and Maintenance Guide along with the LEARN Program CD set. Ann Wellock, a Registered Dietician from The Reading Hospital and Medical Center will deliver the intervention in 2 groups of 20 people that meet weekly for 6 months.
  Interventions: Behavioral: Weight-Centered (LEARN)

INTERVENTIONS:
Behavioral: Wellness-Centered (HUGS) — A health at every size intervention, the HUGS program was conceived and developed in 1987 by Linda Omichinski, Registered Dietitian. HUGS stands for Health focused, Understanding lifestyle, Group supported, and Self-esteem building. It is an integrated approach that promotes healthy eating, active living, and self acceptance regardless of weight. HUGS teaches strategies to recognize and respond to physiological signs of hunger and satiety to determine food intake. The manualized curriculum is accompanied by the books Tailoring Your Tastes and Staying Off of the Diet Roller Coaster which participants will receive in addition to a booklet of handouts. Kelly Bliss, a psychotherapist and fitness professional with 17 years experience in health-centered approaches for weight management, will deliver the intervention in 2 groups of 20 people that meet weekly for 6 months.
  Other Names: Health At Every Size; Intuitive Eating
  Arms: Wellness-Centered
Behavioral: Weight-Centered (LEARN) — The LEARN Program for Weight Management is an evidence-based behavior modification approach to weight loss developed by Dr. Kelly Brownell, Ph.D. Psychologist. LEARN is an acronym that stands for Lifestyle, Exercise, Attitudes, Relationships, and Nutrition. This manualized curriculum shares many principals with the HUGS program in that both emphasize the importance of healthy lifestyle choices and gradual sustainable change. However, the LEARN program makes weight loss an explicit goal and focuses more on food intake levels based on external prescriptions and caloric restriction. Participants in the LEARN program will receive the LEARN Program for Weight Management manual and the LEARN Weight Stabilization and Maintenance Guide along with the LEARN Program CD set. Ann Wellock, a Registered Dietician from The Reading Hospital and Medical Center will deliver the intervention in 2 groups of 20 people that meet weekly for 6 months.
  Other Names: behavior based weight loss program
  Arms: Weight-Centered

SUMMARY:
For over four decades the medical literature has observed a relationship between obesity and poorer health outcomes. The causal mechanisms of these poorer outcomes however are unclear. One assumption that has been supported by correlational data is that increased weight is associated with increased cardiovascular disease (CVD) risk factors (i.e., hypertension, dyslipidemia, and type 2 diabetes). Consequently, obese people are routinely prescribed weight loss programs in order to prevent or control these conditions. Unfortunately, long term weight loss has been met with minimal success for the large majority of people. Furthermore, the data suggesting that weight loss leads to long term health benefits and decreased mortality is limited and contradictory. The purpose of the proposed project is to perform a randomized controlled pilot study comparing the effectiveness of two lifestyle interventions for preventing CVD risk factors (hypertension, dyslipidemia, and type 2 diabetes). The interventions are constitutionally similar; however, the treatment condition is a wellness-focused intervention that teaches healthy living without consideration of weight. The control condition is a traditional curriculum where the prescribed outcome is weight loss. The primary goals of both programs are to reduce hypertension and total cholesterol, and to enhance glucose control. Secondary outcomes of interest are psychological and behavioral in nature (e.g., self-esteem; depressed mood; anxiety; stress; quality of life; dietary habits; and physical activity). We will compare the trajectories of the CVD and psychological/behavioral risk factors for a total period of 24 months (including the time from baseline to the end of the 6-month intervention). Our objectives are to collect data to a) determine whether participants in both programs reduce CVD and psychological/behavioral risk factors at the completion of the 6-month program, and b) compare the persistency of health improvements and rate of relapse at the end of the 18-month follow-up period between the traditional weight loss intervention and the wellness-focused intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 30 to 45 years old (at intervention onset);
2. BMI between 30 and 45
3. Physically inactive
4. Practicing birth control if heterosexually active and pre-menopausal.
5. English speaking

Exclusion Criteria:

1. Current smoker
2. Use of medications known to affect weight/energy expenditure;
3. Pregnant, intending to get pregnant over next two years, or lactating;
4. Recent myocardial infarction (within 6 months);
5. Congestive heart failure
6. Active neoplasms
7. Type 1 and insulin-dependent Type 2 diabetes
8. Cerebrovascular disease
9. Renal disease
10. Cirrhosis
11. Bulimia nervosa
12. Alcohol and/or Substance Abuse
13. Major psychiatric disturbance (suicidality, psychosis, anti-social personality disorder, current manic episode)
14. Prior bariatric surgery
15. Plans to have bariatric surgery over next 2.5 years

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09-25 (Actual); Primary Completion 2011-02-25 (Actual); Study Completion 2011-02-25 (Actual)

PRIMARY OUTCOMES:
Blood Lipids | Baseline, post-intervention, 18-24 months post intervention
  LDL, HDL, Total Cholesterol, Triglycerides (mg/dL)
Blood Pressure | Baseline, post-intervention, 18-24 months post intervention
  Systolic and Diastolic (mmHg)
Fasting Blood Glucose | Baseline, post-intervention, 18-24 months post intervention
  measured in mg/DL
Waist and Hip Circumference | Baseline, post-intervention, 18-24 months post intervention
  measured in inches
Waist-to-Hip ratio | Baseline, post-intervention, 18-24 months post intervention
  waist in inches/hips in inches

SECONDARY OUTCOMES:
Disordered eating attitudes and behaviors | baseline, post intervention, 18-24 months post intervention
  measured using the Eating Disorder Examination-Questionnaire (version 6), Range: 0-6, higher scores indicate worse outcome
Intuitive eating behaviors | baseline, post intervention, 18-24 months post intervention
  Ability to engage in 'adaptive' eating (e.g., recognize internal signs of hunger and satiety) measured the Intuitive Eating Scale. Range: 1-5, higher scores indicate a better outcome
Maladaptive eating behaviors | baseline, post intervention, 18-24 months post intervention
  Measured using the 'emotional eating' and 'uncontrolled eating' eating sub-scales of the Three-Factor Eating Questionnaire -Revised 18, Range: 0-100, higher scores indicate worse outcome
Fruit and vegetable intake | baseline, post intervention, 18-24 months post intervention
  Assessed with the questions: "I eat 2 or more servings of fruit/vegetables on average each day." from the Red Lotus Health and Well-being Questionnaire, Range 0: (none of the time) to 5 (all of the time), higher scores indicate better outcome
Physical activity | baseline, post intervention, 18-24 months post intervention
  Assessed with the question: "I participate in moderately vigorous physical activity for about 30 minutes on average most days of the week." from the Red Lotus Health and Well-being Questionnaire, Range 0: (none of the time) to 5 (all of the time), higher scores indicate better outcome
Self-esteem | baseline, post intervention, 18-24 months post intervention
  measured using the Rosenberg Self-esteem Scale, Range: 0-30, higher scores indicate a better outcome
Overall health and well-being status/Quality of life | baseline, post intervention, 18-24 months post intervention
  measured using the Red Lotus Health and Well-being Questionnaire, Range: 15-75, higher scores indicate a better outcome
Psychological distress | baseline, post intervention, 18-24 months post intervention
  measured using the Depression Anxiety Stress Scale-21, Range: 0-168, higher scores indicate a worse outcome
Dietary habits | baseline, post intervention, 18-24 months post intervention
  Assessment of foods most often consumed, measured using the Dietary Risk Assessment screener, Range 0-125, higher scores indicate higher worse outcome

OTHER OUTCOMES:
Internalized weight stigma (putative mediator and moderator) | baseline, post intervention,18-24 months post intervention
  Degree to which someone personally endorses and adopts negative attitudes about higher weight bodies for themselves. Measured using the Weight Bias Internalization Scale, Range: 1-7, higher scores indicate worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Janell L Mensinger, Ph.D., Principal Investigator — Villanova University
Locations (1):
- The Reading Hospital and Medical Center, West Reading, Pennsylvania, United States

REFERENCES:
- [Result] Mensinger JL, Calogero RM, Stranges S, Tylka TL. A weight-neutral versus weight-loss approach for health promotion in women with high BMI: A randomized-controlled trial. Appetite. 2016 Oct 1;105:364-74. doi: 10.1016/j.appet.2016.06.006. Epub 2016 Jun 8. PMID 27289009
- [Result] Mensinger JL, Calogero RM, Tylka TL. Internalized weight stigma moderates eating behavior outcomes in women with high BMI participating in a healthy living program. Appetite. 2016 Jul 1;102:32-43. doi: 10.1016/j.appet.2016.01.033. Epub 2016 Jan 29. PMID 26829370
- [Result] Mensinger, J. L., & Meadows, A. (2017). Internalized weight stigma mediates and moderates physical activity outcomes during a healthy living program for women with high body mass index. Psychology of Sport and Exercise, 30, 64-72. doi:10.1016/j.psychsport.2017.01.010
- See also: Link to request first publication (main outcomes) from ResearchGate — https://www.researchgate.net/publication/303915874_A_weight-neutral_versus_weight-loss_approach_for_health_promotion_in_women_with_high_BMI_A_randomized-controlled_trial
- See also: Link to request third publication (physical activity mediation and moderation) from ResearchGate — https://www.researchgate.net/publication/313273294_Internalized_weight_stigma_mediates_and_moderates_physical_activity_outcomes_during_a_healthy_living_program_for_women_with_high_body_mass_index